CLINICAL TRIAL: NCT02029989
Title: Can Point-of-care Testing (POCT) and Assistance From Comprehensive Medication Management (CMM) Pharmacists Improve Early Detection and Management of Metabolic Syndrome in Patients Treated With Antipsychotic Medications?
Brief Title: Point-of-Care Testing (POCT) Detection and Management of Metabolic Syndrome in Patients With Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: Medica Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Screening
Other Study IDs: 090M72212
Record Dates: First submitted 2013-09-30; First posted 2014-01-08 (Estimated); Results first posted 2014-05-15 (Estimated); Last update posted 2024-04-04 (Actual); Status verified 2024-04

CONDITIONS: Hyperlipidemia; Diabetes; Hypertension
Keywords: Metabolic Syndrome; Antipsychotics; Schizophrenia; Bipolar Disorder; Diabetes; Dyslipidemia; Hyperlipidemia; Hypertension; Obesity; Medication Therapy Management (MTM); Pharmacist; Comprehensive Medication Management (CMM); Health Disparity; Monitoring; Point of Care Testing; Chronic Persistent Mental Illness
MeSH Terms: conditions — Hyperlipidemias; Diabetes Mellitus; Hypertension; Metabolic Syndrome; Schizophrenia; Bipolar Disorder; Dyslipidemias; Obesity | interventions — Blood Pressure; Heart Rate; Body Mass Index; Carubicin; Medication Therapy Management; myotubularin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Extended Treatment Group (Experimental): Glucose and Lipids and Glycosylated Hemoglobin A1c and Blood Pressure and Heart Rate and Body Mass Index and Waist and Hip Circumference and Comprehensive Medication Management
  Interventions: Device: Glucose and lipids; Device: Glycosylated Hemoglobin A1c; Device: Blood Pressure and Heart Rate; Device: Body mass index; Device: Waist and Hip circumference; Behavioral: Comprehensive Medication Management
- Usual Treatment Group (Active Comparator): Glucose and Lipids and Glycosylated Hemoglobin A1c and Blood Pressure and Heart Rate and Body Mass Index and Waist and Hip Circumference
  Interventions: Device: Glucose and lipids; Device: Glycosylated Hemoglobin A1c; Device: Blood Pressure and Heart Rate; Device: Body mass index; Device: Waist and Hip circumference

INTERVENTIONS:
Device: Glucose and lipids — Point-of-care (POCT) screening for diabetes and dyslipidemia.
  Glucose and Lipids
  Other Names: Cholestech LDX ® by Inverness Medical www.cholestech.com
Device: Glycosylated Hemoglobin A1c — Point-of-care (POCT) screening for diabetes
  Glycosylated Hemoglobin A1c
  Other Names: A1c Now® by Bayer HealthCare
Device: Blood Pressure and Heart Rate — Point-of-care (POCT) screening for hypertension
  Blood Pressure and Heart Rate
  Other Names: Omron ® Ultra Premium blood pressure monitor Model HEM-790IT
Device: Body mass index — Height and weight measurement used to calculate BMI = Mass(kg)/(height (m))squared
  Other Names: HealthOMeter® 500KL
Device: Waist and Hip circumference — Measurement for Central Obesity
  Waist and Hip circumference
  Other Names: QM2000 Circumference measuring tape
Behavioral: Comprehensive Medication Management — Defined at http://www.pcpcc.org/guide/patient-health-through-medication-management
  Other Names: CMM, Medication Therapy Management, MTM
  Arms: Extended Treatment Group

SUMMARY:
The study was a 12-month, multi-centered, quasi-experimental design to assess point-of-care (POCT) screening/monitoring of subjects on antipsychotic agents for metabolic syndrome. Subjects were also randomized to either an Extended Treatment Group (ETG) defined by receiving comprehensive medication management (CMM) pharmacist interventions or a Usual Treatment Group (UTG) receiving no CMM interventions. All subjects were recruited from three community mental health clinic settings in Minnesota.

DETAILED DESCRIPTION:
It is well recognized that patients on antipsychotic agents with mental illness continue to be affected by a severe health disparity due to lack of adequate metabolic monitoring.1-7 A major healthcare concern is the life-expectancy decrease of ~25 years for patients with illnesses such as schizophrenia as compared with the general population. Equally concerning is that patients with severe persistent mental illness (SPMI) continue to have inadequate integration of care between psychiatry and medicine. Because of the difficulty getting patients to primary care or hospital based laboratories, the use of capillary blood, point-of-care tests (POCT) to monitor glucose and lipids in addition to vital signs and other anthropometric measurements in community mental health centers might prove beneficial. It is highly likely that this advanced level of screening in the mental health setting may lead to identifying new metabolic abnormalities or improved treatment with careful monitoring of previously diagnosed metabolic syndrome, diabetes, and/or hypertension in antipsychotic treated patients. It is hypothesized that if metabolic abnormalities are identified; then providing pharmacist CMM consultative services would reduce medication related problems by improving medication adherence, coordination of care between psychiatry and primary care, and outcomes in metabolic indices.

ELIGIBILITY:
Inclusion Criteria:

* English speaking
* Age 18-64
* Competent to understand and make medical choices independently

Exclusion Criteria:

* Currently or previously seen by a CMM pharmacist

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 121 (Actual)
Dates: Start 2010-02; Primary Completion 2012-02 (Actual); Study Completion 2012-02 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Human Development Center, Duluth, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schneiderhan ME, Shuster SM, Davey CS. Twelve-month prospective randomized study of pharmacists utilizing point-of-care testing for metabolic syndrome and related conditions in subjects prescribed antipsychotics. Prim Care Companion CNS Disord. 2014 Oct 30;16(5):10.4088/PCC.14m01669. doi: 10.4088/PCC.14m01669. eCollection 2014. PMID 25667811
- [Result] Schneiderhan ME, Li X. Observed Sex Differences in Cardiometabolic Indices in Patients on Antipsychotics: Secondary Analyses of a 12-Month Multicenter, Randomized, Controlled Trial. Prim Care Companion CNS Disord. 2021 Apr 8;23(2):19m02493. doi: 10.4088/PCC.19m02493. PMID 34000112

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at three community mental health sites in Minnesota site (Human Development Center - Duluth, MN; Range Mental Health Center - Hibbing, MN; Family Life Mental Health Center - Coon Rapids, MN; with subjects assigned to receive either pharmacist CMM services (PCS) or no pharmacist CMM services (NCS)/Control Group.
Groups:
- Pharmacist Comprehensive Medication Management Service (PCS): Glucose and Lipids and Glycosylated Hemoglobin A1c and Blood Pressure and Heart Rate and Body Mass Index and Waist and Hip Circumference and Comprehensive Medication Management
  Cholestech LDX ®: Point-of-care (POCT) screening for diabetes and dyslipidemia.
  Glucose and Lipids
  A1c Now®: Point-of-care (POCT) screening for diabetes
  Glycosylated Hemoglobin A1c
  Omron ® Ultra Premium blood pressure monitor Model HEM-790IT: Point-of-care (POCT) screening for hypertension
  Blood Pressure and Heart Rate
  HealthOMeter® 500KL: Height and weight measurement used to calculate BMI = Mass(kg)/(height (m))squared
  QM2000 Circumference measuring tape: Measurement for Central Obesity
  Waist and Hip circumference
  Comprehensive Medication Management: Defined at http://www.pcpcc.org/guide/patient-health-through-medication-management
- No Comprehensive Medication Management Services (NCS): Glucose and Lipids and Glycosylated Hemoglobin A1c and Blood Pressure and Heart Rate and Body Mass Index and Waist and Hip Circumference
  Cholestech LDX ®: Point-of-care (POCT) screening for diabetes and dyslipidemia.
  Glucose and Lipids
  A1c Now®: Point-of-care (POCT) screening for diabetes
  Glycosylated Hemoglobin A1c
  Omron ® Ultra Premium blood pressure monitor Model HEM-790IT: Point-of-care (POCT) screening for hypertension
  Blood Pressure and Heart Rate
  HealthOMeter® 500KL: Height and weight measurement used to calculate BMI = Mass(kg)/(height (m))squared
  QM2000 Circumference measuring tape: Measurement for Central Obesity
  Waist and Hip circumference
Period: Overall Study
Arm/Group | Pharmacist Comprehensive Medication Management Service (PCS) | No Comprehensive Medication Management Services (NCS)
Started | 61 (A subject was given the same ID# as withdrawn subject (ID # counted twice) causing N=61 discrepancy.) | 60
Completed | 45 | 49
Not Completed | 16 | 11
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Withdrawal: Fear of needles | 1 | 0
Not completed — Change of location | 2 | 3
Not completed — Physician Decision | 2 | 0
Not completed — Lost to Follow-up | 9 | 7
Not completed — Death | 0 | 1
Not completed — Protocol Violation | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Pharmacist Comprehensive Medication Management Service (PCS) | No Comprehensive Medication Management Services (NCS) | Total
Number analyzed (Participants) | 60 | 60 | 120
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.32 (11.95) | 43.5 (10.62) | 42.9 (11.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 36 | 35 | 71
  Male | 24 | 25 | 49
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1
  Asian | 1 | 1 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 4 | 1 | 5
  White | 51 | 53 | 104
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 4 | 8
Subjects with Metabolic Syndrome based on Point of Care analyses [Number; unit: participants] — Metabolic syndrome was identified in 71.2% of the NCS group and in 85.2% of the PCS group. Data was not available for 7 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 46 | 42 | 88
Abdominal Obesity [Number; unit: participants] — Waist Circumference Risk (Males: > 40 inches, Females: > 35 inches) was 86.4% in the NCS group and 87.7% in the PCS Group. Data was not available for 4 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 50 | 51 | 101
Total Cholesterol Risk [Number; unit: participants] — Risk is defined as greater than 200 mg/dL was 41.7% in the NCS group and 38.6% in the PCS group. Data was not available for 3 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 22 | 25 | 47
Low Density Lipoprotein (LDL) Risk [Number; unit: participants] — Risk is defined as greater than 130 mg/dL was 24.5% in the NCS group and 25.5% in the PCS group. Data was not available for 20 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 13 | 12 | 25
Triglyceride Risk [Number; unit: participants] — Risk is defined as greater than 150 mg/dL was 54.2% in the NCS group and 42.1% in the PCS group. Data was not available for 4 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 24 | 32 | 56
High Density Lipoprotein (HDL) Risk [Number; unit: participants] — Risk is defined as: Males < 40 mg/dL; Females < 50 mg/dL was 75% in the NCS group and 73.3% in the PCS group. Data was not available for 7 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 44 | 45 | 89
Hypertension Risk [Number; unit: participants] — Risk is defined as blood pressures greater than 130 mmHg systolic and/or greater than 85 mmHg diastolic was 48.1% in the NCS group and 51.9% in the PCS group. Data was not available for 2 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 27 | 25 | 52
Diabetes Risk [Number; unit: participants] — Risk is defined as glycosylated hemoglobin A1c greater or equal to 6.5% was found in 10.3% of the NCS group and 12.5% of the PCS group. Data was not available for 6 subjects. This explains why the sum of this baseline measure does not equal the overall baseline participants.
  participants | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Metabolic Syndrome (MetS)
Description: compare test results in subjects between the PCS and NCS groups, with or without pre-existing MetS and/or related metabolic conditions at baseline
Time Frame: Baseline
Measure: Number; unit: percentage of participants
Arm/Group | Pharmacist Comprehensive Medication Management Service (PCS) | No Comprehensive Medication Management Services (NCS)
Number analyzed (Participants) | 60 | 60
percentage of participants | 85.2 | 71.2

ADVERSE EVENTS:
Arm/Group | Pharmacist Comprehensive Medication Management Service (PCS) | No Comprehensive Medication Management Services (NCS)
Serious Adverse Events (participants affected / at risk) | 0/60 | 0/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60

LIMITATIONS AND CAVEATS:
Limitations include: 1) Short time duration to achieve metabolic outcome goals, 2) Smaller than anticipated sample size, 3) High number of subjects lost to follow up after 12-months.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No